CLINICAL TRIAL: NCT02558478
Title: Identification of New Genes Implicated in Rare Neurosensory Diseases by Whole Exome Sequencing
Acronym: GEN-NEUROSENS
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: University Hospital, Strasbourg, France (Other)
Responsible Party: Sponsor
Other Study IDs: 5885
Record Dates: First submitted 2015-09-11; First posted 2015-09-24 (Estimated); Last update posted 2016-12-07 (Estimated); Status verified 2016-12

CONDITIONS: Neurosensory Diseases; Retinopathy; Hearing Loss
Keywords: Whole exome sequencing
MeSH Terms: conditions — Retinal Diseases; Hearing Loss | interventions — Blood Specimen Collection

STUDY DESIGN:
Observational Model: Family Based
Biospecimen Retention: Samples With DNA — DNA Fibroblasts
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Genetic: blood sampling

SUMMARY:
Next Generation Sequencing (NGS) strategy is a powerful tool to identify genes implicated in very rare diseases for which the previous genetic explorations remain negative to date. The aim of this project is based on groups of patients with original clinical phenotypes including neurosensory impairment without genetic cause identified to date. The investigators will study these families using whole exome sequencing to potentially identify new genes and new underlying biological pathways involved in neurosensory diseases.

ELIGIBILITY:
Inclusion Criteria:

* Original phenotype with neurosensory diseases
* Written, informed consent obtained

Exclusion Criteria:

* Refusal to participate at the study
* Prior inclusion in a similar study (NGS)

Ages: 28 Days to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: This project focuses on families with unsual phenotypes who have sensorineural disease with retinal degeneration AND/OR deafness. Our first hypothesis is that these clinical entities are associated with new genes not described to date. However, it is impossible to exclude at this stage an allelic variability (mutations in genes already known but with an unusual phenotype) or mutations in genes implicated in neurosensory diseases but not detected by prior exploration. These situations illustrate the problem of genetic complexity and difficulty of the phenotype correlations - genotype.
Sampling Method: Non-Probability Sample
Enrollment: 39 (Estimated)
Dates: Start 2015-09; Primary Completion 2018-09 (Estimated); Study Completion 2018-09 (Estimated)

PRIMARY OUTCOMES:
Whole exome sequencing data | 21 months

CONTACTS AND LOCATIONS:
Overall Officials: Sophie SCHEIDECKER, MD, Principal Investigator — Hôpitaux Universitaires de Strasbourg
Locations (1):
- LABORATOIRE DE CYTOGENETIQUE, Hôpitaux Universitaires de Strasbourg, Strasbourg, France